CLINICAL TRIAL: NCT03373929
Title: Suture Mediated Septal Defect Closure/Repair Evaluation of the NobleStitch EL System
Brief Title: Stitch Closure of PFO and Septal Repair
Acronym: STITCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HeartStitch.Com (Industry)
Responsible Party: Principal Investigator, James Thompson, MD, Interventional Cardiologist, HeartStitch.Com
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-2871
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Foramen Ovale, Patent; Septal Defect, Atrial; Septal Defect, Heart
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Septal Defects, Atrial; Heart Septal Defects

STUDY DESIGN:
Intervention Model Description: Non-randomized, single-center, observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PFO Closure Rate (Other): Evaluate closure rate of clinically relevant septal defects including PFO, ASD (less than 1 cm with redundant septal tissue), trans septal puncture sites, repair of ASA (when an appropriate PFO or small ASD defect is present) and rate of recurrent neurologic embolic event in patients with cryptogenic stroke and PFO
  Interventions: Device: PFO Closure Rate; Device: Published PFO Device Closure
- Published PFO Device Closure (Other): Compare PFO closure rate and safety of closure of septal occluders in published PFO clinical trials.
  Interventions: Device: PFO Closure Rate; Device: Published PFO Device Closure

INTERVENTIONS:
Device: PFO Closure Rate — Suture Mediated PFO Closure and Septal Repair
Device: Published PFO Device Closure — Suture Mediated PFO Closure and Septal Repair

SUMMARY:
The purpose of the STITCH study is to evaluate closure rates of clinically relevant septal defects, including patent foramen ovale (PFO), Atrial Septal Defects (ASD - less than 1 cm with redundant septal tissue), trans septal puncture sites, repair of Atrial Septal Aneurysm (ASA) and rate of recurrent neurologic embolic events in patients with cryptogenic stroke and PFO.

ELIGIBILITY:
Inclusion Criteria:

* PFO
* ASD (less than 1 cm with redundant septal tissue)
* Trans Septal Puncture Sites
* ASA (when an appropriate PFO or small ASD defect is present)
* Stroke
* Trans ischemic Attack (TIA)
* Platypnea Orthodeoxia Syndrome
* Decompression Illness

Exclusion Criteria:

* Patients under 18 and over 65
* Patients who are not fluent in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-11-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Closure Rates of PFO and ASD | 12 months
  Saline Contrast Echo

SECONDARY OUTCOMES:
Recurrent Stroke Rate | 4-6 weeks, 6 months, 1 year and annually up to five years
  Rate of which Patient Experiences Recurrent Stroke

OTHER OUTCOMES:
Migraine | 4-6 weeks, 6 months, 1 year and annually up to five years
  Rate of Patients who have Experienced Improvement in Migraine

CONTACTS AND LOCATIONS:
Overall Officials: James Thompson, MD, Principal Investigator — Inova Cardiovascular Institute
Locations (1):
- Inova Cardiovascular Institute, Falls Church, Virginia, United States